CLINICAL TRIAL: NCT00295087
Title: X-Chromosome Inactivation Status and Premature Ovarian Failure
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 0511043
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Premature Ovarian Failure
Keywords: Premature Ovarian Failure; X-Chromosome Inactivation
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA that is extracted from the blood specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Women who are affected with premature ovarian failure will exhibit skewed X-chromosome inactivation patterns compared to women with normal menstrual function (as defined by being pregnant), indicating a possible X-chromosome defect.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) affects approximately 1% of women. For most women a cause is not found, but structural abnormalities of the X-chromosome commonly lead to POF, suggesting genes on the X-chromosome are necessary for normal ovarian function. It is known that certain gene mutations on the X-chromosome can lead to changes in the normal random pattern of X-chromosome inactivation in females.

We propose to study X-inactivation patterns in a cohort of women with idiopathic POF, and compare their pattern to a mean age-matched cohort of women with normal menstrual function.

We hypothesize that some women with POF will show skewed X-inactivation, suggesting a mutation on the X-chromosome as the etiology of their POF.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with POF.
* A chromosomal analysis must have been performed to evaluate X-chromosomal abnormalities, and the results are known to be normal.

Exclusion Criteria:

* Patients who have a known etiology for their POF and/or an inability to obtain karyotype results for these patients or unknown X-chromosome abnormalities.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will include women diagnosed with POF through clinics. Women diagnosed with POF may also inquire about this study through the Clinical Trials website.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2005-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Skewed X-Inactivation appears increased in women with Premature Ovarian Failure | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: W. Allen Hogge, MD, Principal Investigator — University of Pittsburgh and Magee-Womens Hospital
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States